CLINICAL TRIAL: NCT07138846
Title: A Randomized, Double-blind, Multi-center, Phase III Study of MRG004A Plus Best Supportive Care Versus Placebo and Best Supportive Care in the Treatment of Patients With Advanced Pancreatic Cancer
Brief Title: A Study Comparing MRG004A Plus Best Supportive Care Versus Placebo and Best Supportive Care in the Treatment of Patients With Advanced Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRG004A-002
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Advanced Pancreatic Cancer
Keywords: MRG004A; Best Supportive Care; Placebo Controlled; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Interventions administered to this arm include MRG004A, which is the investigational drug product, plus best supportive care, including but not limited to pain management, nutrition support, and psychological therapy
  Interventions: Drug: MRG004A plus best supportive care
- Control Arm (Placebo Comparator): Placebo plus best supportive care, the definition of best supportive care is the same as that in the experiment arm
  Interventions: Drug: Placebo plus best supportive care

INTERVENTIONS:
Drug: MRG004A plus best supportive care — MRG004A will be administrated as specified in the protocol.
  Arms: Experimental Arm
Drug: Placebo plus best supportive care — Placebo will be administrated as specified in the protocol, following the same dose regimen as MRG004A.
  Arms: Control Arm

SUMMARY:
This is a randomized, double-blind, multi-center, phase III study to evaluate the efficacy and safety, pharmacokinetic profile and immunogenicity of MRG004A in patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the informed consent form and follow the requirements specified in the protocol.
* Patients with histologically and cytologically confirmed locally advanced or metastatic pancreatic cancer, including adenocarcinoma, who have failed at least prior systemic therapies including gemcitabine and fluorouracil.
* Patients must have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
* The score of ECOG for performance status is 0 to 2.
* Organ functions and coagulation function must meet the basic requirements.
* Patients with childbearing potential must use effective contraception during the treatment and for 6 months after the last dose of treatment.

Exclusion Criteria:

* History of other primary malignant tumors
* Active metastasis to brain or meninges
* Active acute or chronic inflammatory skin disease, history of Steven-Johnson syndromes
* History of active or chronic corneal and conjunctival diseases, or other clinically significant ocular diseases that affect the ophthalmic monitoring of the investigational drug
* Received certain anti-tumor therapies or strong CYP3A4 inhibitors and have not complete the wash-out period, or have not fully recovered from major surgery
* AEs due to prior anti-tumor therapy(ies) that have not resolved to ≤Grade 1 per CTCAE v5.0
* Presence of ≥Grade 2 peripheral neuropathy per CTCAE v5.0
* Poorly controlled pleural and peritoneal effusion or pericardial effusion
* Severe cardiac dysfunction within 6 months before enrollment
* History of ventricular tachycardia, or torsade des pointes
* Uncontrolled or poorly controlled hypertension
* Compression fractures of the spine that have not been treated with surgery and/or radiation therapy, or have not been stable within 2 weeks before randomization
* Pulmonary embolism or deep vein thrombosis within 3 months prior to the first dose of study drug.
* Patients with high risk of bleeding per investigator's judgement.
* Patients who have active infection including but not limited to hepatitis B, hepatitis C, AIDS, or syphilis.
* Active uncontrolled bacterial, viral, fungal, rickettsial, or parasitic infection.
* Moderate to severe dyspnea at rest, severe primary lung disease, interstitial lung disease, or pneumonia.
* Uncontrolled pain due to cancer
* Active or history of autoimmune disease that requiring systemic hormone therapy
* History of hypersensitivity to any component of the investigational product.
* Other situations that are not suitable to participate a clinical trial per investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Baseline to study completion (up to 24 months)
  OS is defined as the duration from the start of treatment to death of any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Baseline to study completion (up to 24 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Objective Response Rate (ORR) | Baseline to study completion (up to 24 months)
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed according to RECIST v1.1.
Disease Control Rate (DCR) | Baseline to study completion (up to 24 months)
  DCR is defined as the proportion of subjects achieving CR, PR, and stable disease (SD) after treatment.
Duration of Response (DOR) | Baseline to study completion (up to 24 months)
  The time interval between the date of the earliest qualifying response and the date of disease progression or death for any cause, whichever occurs earlier.
Immunogenicity (ADA) | Baseline to 14 days after the last dose.
  The proportion of patients with positive ADA results.
Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Serious Adverse Events (SAEs) | Baseline to 30 days after the last dose of study treatment
  Adverse events that are fatal, life-threatening, or result in hospitalization or prolonged hospitalization, persistent or significant disability/incapacity/substantial disruption of the ability to lead a normal life, congenital anomaly/birth defect or major medical events or reactions

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No